CLINICAL TRIAL: NCT05222672
Title: Electrical and Mechanical Activation in PAcing The His Bundle Conduction sYstem: EMPATHY Study
Brief Title: Electrical and Mechanical Activation in PAcing The His Bundle Conduction sYstem
Acronym: EMPATHY
Status: Completed | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Matteo Bertini, Principal Investigator, University Hospital of Ferrara
Other Study IDs: CE-AVEC 457/2021/Oss/AOUFe
Record Dates: First submitted 2022-01-17; First posted 2022-02-03 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Pacemaker DDD; His Bundle Pacing; Right Ventricular Pacing
Keywords: 3D mapping system; Myocardial work; Mechanical dyssynchrony; 12-lead Electrocardiogram; Speckle-tracking echocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: His Bundle Pacing — Pacing of the His bundle

SUMMARY:
In recent years, the finding of long-term deleterious effects of right ventricular pacing (RVP) has led to an ongoing search for alternative pacing sites such as His bundle stimulation. The depolarization of the ventricles through the His-Purkinje cardiac conduction system seems to represent an ideal physiological approach to ventricular pacing, capable of engaging the normal conduction pathways and determining synchronous ventricular activation. However, there are still no clinical studies that have evaluated the electromechanical functions of the left ventricle with His bundle pacing (HBP) identified after electroanatomical reconstruction with 3D mapping system. Investigators aimed to compare the electromechanical effects on left ventricle of HBP, compared to RVP stimulation and to spontaneous rhythm of each patient.

DETAILED DESCRIPTION:
Patients with indication for permanent pacemaker implantation were included in the study. The stimulation lead was positioned at the level of the His bundle after complete electroanatomical reconstruction of the atrium and right ventricle with 3D mapping system; a second backup lead was eventually placed in the right ventricle. Within 24 hours after implantation, each patient underwent 12-lead ECG and a complete echocardiographic examination in the different pacing modalities (HBP, RVP and patient's spontaneous rhythm) focused on the evaluation of biventricular systo-diastolic function, speckle-tracking and myocardial work of the left ventricle.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication of class I or class IIa for permanent pacemaker implantation, in accordance with the guidelines of the European Society of Cardiology on cardiac pacing
* Age ≥ 18 years
* Written consent

Exclusion Criteria:

* Patients unable to express informed consent
* Pregnancy
* Severe mitro-aortic valve disease
* Left ventricular ejection fraction ≤ 35%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over the age of 18 years with indication for permanent pacemaker implantation.
Sampling Method: Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Evaluate the electrocardiographic differences of HBP, obtained by electroanatomical reconstruction with 3D mapping system, compared to the RVP and the patient's spontaneous rhythm. | 24 hours after implantation
  Measurement of QRS width (msec) in 12-lead electrocardiogram
Evaluate the echocardiographic differences of HBP, obtained by electroanatomical reconstruction with 3D mapping system, compared to the RVP and the patient's spontaneous rhythm. | 24 hours after implantation
  Transthoracic echocardiogram measurement such as left ventricular systolic function (%), left ventricular Global Longitudinal Strain (GLS %), tissue doppler and severity of any valve disease

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Bertini, MD, PhD, Principal Investigator — Università degli Studi di Ferrara
Locations (1):
- Azienda Ospedaliero-Universitaria di Ferrara, Ferrara, Italy

REFERENCES:
- [Result] Malagu M, Vitali F, Massafra RF, Cardelli LS, Pavasini R, Guardigli G, Rapezzi C, Bertini M. Three-Dimensional Electro-Anatomical Mapping and Myocardial Work Performance during Spontaneous Rhythm, His Bundle Pacing and Right Ventricular Pacing: The EMPATHY Study. J Cardiovasc Dev Dis. 2022 Nov 2;9(11):377. doi: 10.3390/jcdd9110377. PMID 36354776